CLINICAL TRIAL: NCT01890239
Title: Improving End-of-life Care in Acute Geriatric Hospital Wards Using the Care Programme for the Last Days of Life: a Cluster Randomized Controlled Trial
Brief Title: The Effectiveness of the Care Programme for the Last Days of Life
Acronym: PLaDays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: End-of-Life Research Group (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other); KU Leuven (Other); Amsterdam UMC, location VUmc (Other); University Ghent (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Tinne Smets, Doctoral reseracher, End-of-Life Research Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B143201213985
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Older Patients Dying in Acute Geriatric Hospital Wards

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Programme for the Last Days of Life (Experimental): The Care Programme for the Last Days of Life will be implemented in the acute geriatric hospital wards randomized to the experimental group. Subsequently, older patients hospitalized in one of these experimental wards and for who the multidisciplinary team has decided that he or she has entered the dying phase, will benefit from this Care Programme.
  Interventions: Other: Care Programme for the Last Days of Life
- Usual care (No Intervention): Care will be provided as usual, also for patients who have entered the dying phase.

INTERVENTIONS:
Other: Care Programme for the Last Days of Life — The Care Programme essentially aims to raise awareness among geriatric health care staff of the importance for improving end-of-life care and to prepare them for a change in end-of-life care, to train staff in delivering good end-of-life care with the support of a multi-professional document called the Care Guide for the Last Days of Life, to support dying geriatric patients with the Care Guide for the Last days of Life, to regularly evaluate the delivered end-of-life care and support and to further educate the staff in delivering optimal end-of-life care. The Care Programme consists of the following documents: (1) the Care Guide for the Last Days of Life, (2) supportive documentation and (3) an implementation guide.
  Arms: Care Programme for the Last Days of Life

SUMMARY:
BACKGROUND Demographic trends coupled with a rise in chronic diseases mean that the population of patients requiring palliative and end-of-life care is ageing. Due to the ageing population palliative care for older people has been identified as one of the worldwide public health priorities. A majority of elderly patients die in hospital. Studies from the United Kingdom and other countries have shown that many older persons dying in hospital experience suboptimal care. The Care Programme for the Last Days of Life has been developed to improve the quality of end-of-life care in acute geriatric hospital wards. The programme is based on existing end-of-life care programmes but modeled to the acute geriatric care setting. There is a lack of evidence of the effectiveness of end-of-life care programmes and the effects that may be achieved in patients dying in an acute geriatric hospital setting are unknown. The aim of this study is to evaluate the effectiveness of the Care Programme for the Last Days of Life in improving the quality of care and quality of life during the last 48 hours of life of patients dying in acute geriatric hospital wards in Flanders as compared to usual care.

METHODS In order to contribute substantially to the increase of evidence for the effect of the Care Programme for the Last Days of Life in patients dying in acute geriatric hospital wards, a cluster randomized controlled trial will be conducted. Ten hospitals with one or more acute geriatric wards will conduct a one-year baseline assessment during which care will be provided as usual. For each patient dying in the ward, a questionnaire will be filled in by a nurse, a physician and a family carer. At the end of the baseline assessment hospitals will be randomized to receive intervention (implementation of the Care Programme) or no intervention. Subsequently, the Care Programme will be implemented in the intervention hospitals over a six-month period. A one-year post-intervention assessment will be performed immediately after the baseline assessment in the control hospitals and after the implementation period in the intervention hospitals. Primary outcomes are symptom frequency and symptom burden of patients in the last 48 hours of life.

DISCUSSION This will be the first cluster randomized controlled trial to evaluate the effect of the Care Programme for the Last Days of Life for the acute geriatric hospital setting. The results will enable us to evaluate whether implementation of the Care Programme has positive effects on end-of-life care during the last days of life in this patient population and which components of the Care Programme contribute to improving the quality of end-of-life care.

ELIGIBILITY:
The inclusion criteria of the hospitals in the trial are:

* the cluster or hospital has one or more acute geriatric wards
* the medical and nursing head of one or more acute geriatric wards per hospital give consent for participation in the study

The inclusion criteria of patients are:

* those dying in the acute geriatric ward between October 2012 and March 2015
* those that having been hospitalized for more than 48 hours
* those having given informed consent at admission for the use of their personal information from medical or nursing records for the purposes of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The effect of implementation of the Care Programme for the Last Days of Life on the quality of dying in acute geriatric hospital wards: the patient's symptom frequency and symptom burden evaluated by the SM-EOLD and CAD-EOLD | within 3 months after a patient's death
  Using a cluster randomized controlled trail with randomized assignment to the intervention or control group, the effect of the Care Programme on the quality of dying is evaluated with the SM-EOLD and CAD-EOLD

SECONDARY OUTCOMES:
The quality of care during the last three days of life as perceived by nurses, i.e. physical symptoms, emotional, psychological and spiritual/existential needs and provision of information and support measured using the POS | within 3 months after a patient's death
The quality of care during the last 48 hours of life as perceived by family carers, i.e. satisfaction with the care provided to the patient during the last 48 hours of life measured using the EOLD-SWC | within 3 months after a patient's death
The content of care during the last 48 hours of life, i.e. the goal of treatment, medical and nursing interventions, medication policy | within 3 months after a patient's death
The communication among clinical staff, i.e. informing the family physician about the impending death | within 3 months after a patient's death
The communication between clinical staff and patients and/or family carers, i.e. the perception of communication with the physician during the dying phase by family carers measured using the FPPFC | within 3 months after a patient's death
The level of bereavement of family carers after the death of the patient measured using the PGD scale | within 3 months after a patient's death

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (9):
  - St Jan Brugge, Bruges
  - St Lucas Brugge, Bruges
  - AZ Sint Blasius, Dendermonde
  - Jessa Ziekenhuis Hasselt, Hasselt
  - Sint Jozefskliniek Izegem, Izegem
  - AZ Lokeren, Lokeren
  - H. Hartziekenhuis Menen, Menen
  - Sin Rembertziekenhuis Torhout, Torhout
  - Sint Augustinuskliniek Veurne, Veurne

REFERENCES:
- [Derived] Beernaert K, Smets T, Cohen J, Verhofstede R, Costantini M, Eecloo K, Van Den Noortgate N, Deliens L. Improving comfort around dying in elderly people: a cluster randomised controlled trial. Lancet. 2017 Jul 8;390(10090):125-134. doi: 10.1016/S0140-6736(17)31265-5. Epub 2017 May 16. PMID 28526493
- [Derived] Verhofstede R, Smets T, Cohen J, Costantini M, Van Den Noortgate N, Deliens L. Improving end-of-life care in acute geriatric hospital wards using the Care Programme for the Last Days of Life: study protocol for a phase 3 cluster randomized controlled trial. BMC Geriatr. 2015 Feb 22;15:13. doi: 10.1186/s12877-015-0010-7. PMID 25887959